CLINICAL TRIAL: NCT06244277
Title: Research on High-efficiency of Treatment of Adolescent Sleep Disorders Technology and Sleeping Pills Withdrawal
Brief Title: Chinese Medicine Treatment of Adolescent Sleep Disorders and Sleeping Pills Withdrawal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-850
Record Dates: First submitted 2024-01-15; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Traditional Chinese Medicine; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese medicine group (Experimental): Participants received Suanzaoren Decoction and Huanglian Wendan Decoction orally twice daily for 4 weeks. Subjects who had previously taken Western medicine hypnotics continued to take them, and those who did not take them did not add Western medicine hypnotics.
  Interventions: Drug: Suanzaoren Decoction and Huanglian Wendan Decoction
- Western medicine group (Active Comparator): Participants received cognitive behavioral therapy, if for various reasons can not accept cognitive behavioral therapy, or have received cognitive behavioral therapy is not effective, according to the doctor to consider drug treatment, taking Zolpidem Tartrate Tablets 0.25mg/kg, the maximum dose was 10mg / day ; according to the doctor 's clinical consideration, anxiety and depression drugs can be added. For patients under 18 years of age, under the careful consideration of the doctor for drug treatment, taking Zolpidem tablets, 10mg / day
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Suanzaoren Decoction and Huanglian Wendan Decoction — Twice daily. Chinese herbal medicine includes: includes: 25 grams of Suanzaoren, 10 grams of chuanxiong, 30 grams of fushen, 10 grams of Polygala tenuifolia, 10 grams of Pinellia ternata, 12 grams of tangerine peel, 15 grams of Zhuru, 30 grams of forged keel, 30 grams of forged oyster,10 grams of aurantii fructus, 6 grams of coptis chinensis, 30 grams of Albizzia bark.Add or subtract Chinese herbal medicine according to the different clinical manifestations of each patient.
  Arms: Chinese medicine group
Drug: Zolpidem — Zolpidem 10Mg Tab 10mg tablet once daily
  Arms: Western medicine group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of traditional Chinese medicine in the treatment of adolescent sleep disorders and the effect of sleeping pills withdrawal.

DETAILED DESCRIPTION:
All subjects giving written informed consent. In this multicenter,controlled, prospective cohort study, the outpatient and inpatient adolescent sleep disorder patients' baseline demographic data were collected, including age, gender, education background, and medication history. Venous blood samples were collected and sent to laboratory test for blood routine, and blood biochemistry at Baseline and Week 4. The Pittsburgh sleep quality index (PSQI) was used to assess the patients' sleep quality at baseline, month 1, month 3 and month 6. Objective sleep quality data is assessed by wearing a Sleep wearable devices. The classic Morningness-Eveningness Questionnaire and wearable devices was used to assess the patients' chronotype at baseline and week 4.Subjects who visit the TCM clinic of this project received Suanzaoren Decoction and Huanglian Wendan Decoction and other decoctions orally twice daily for 4 weeks. Add or subtract Chinese herbal medicine according to the different clinical manifestations of each patient. Subjects from TCM clinic who had previously taken Western medicine hypnotics continued taking them, and for those who had not taken before, Western medicine hypnotics shall not be given/prescribed. Subjects who visit the Western medicine clinic of this project received cognitive behavioral therapy, if for various reasons can not accept cognitive behavioral therapy, or have received cognitive behavioral therapy is not effective, according to the doctor to consider drug treatment, taking Zolpidem Tartrate Tablets 0.25mg/kg, the maximum dose was 10mg / day ; according to the doctor 's clinical consideration, anxiety and depression drugs can be added. For patients under 18 years of age, under the careful consideration of the doctor for drug treatment, taking oxazepam tablets, 3.75-15mg / day, if necessary, signed informed consent of clinical medication. Adverse reactions were closely monitored during medication.The participants will have a follow-up visit every two weeks, and the prescription would be adjusted according to the condition of illness.Cessation rate of Western medicine hypnotics was assessed at Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or inpatients.
* It meet the diagnostic criteria of ' International Classification of Sleep Disorders, Third Edition ' ( ICSD-3 )..
* Informed consent, voluntary participation in the study.

Exclusion Criteria:

* Sleep disorders are caused by systemic diseases such as body pain, fever, cough, surgery and external environmental interference.Sleep apnea syndrome leads to insomnia.
* Severe depression, suicidal tendency or having committed suicide.
* Pregnant and lactating women.
* It has serious primary heart, liver, lung, kidney, blood or serious diseases affecting its survival, such as: tumor or AIDS, SCR > 1.5n (n is the upper limit of normal value), ALT > 2n (n is the upper limit of normal value), WBC < 3.0 × 109 / L;
* Those who cannot give full informed consent due to mental disorders.
* According to the researcher's judgment, other situations that are not suitable for the group, such as the change of working environment.
* Subjects who are participating in other clinical studies.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the total score of the Pittsburgh sleep quality index (PSQI) at Month 1 | Baseline and Month 1
  The Pittsburgh sleep quality index (PSQI) is a validated,self-reported instrument assessing the sleep quality over the past 4 week period. Possible scores range from 0(the best sleep quality) to 21(the worst possible sleep) quality).The higher the score of PSQI, the worse the sleep quality. Change=(Month 1 Score-Baseline Score)
Insomnia severity index ( ISI ) score reduction rate at Month 1 | Month 1
  Insomnia severity index ( ISI ) is to assess the nature and symptoms of sleep disorders in subjects. Score reduction rate of Insomnia severity index ( ISI )=(Baseline number-Month 1number)/Baseline number of participants

SECONDARY OUTCOMES:
Cessation rate of Western medicine hypnotics at Month 6 | Month 6
  Cessation is defined as an absence of any Western medicine hypnotics that was sustained for 3 consecutive months or more. Cessation rate of Western medicine hypnotics=(Month 6 number-Baseline number)/Baseline number of Participants use Western medicine hypnotics.
Athens Insomnia Scale ( AIS ) score at Month 1 | Baseline and Month 1
  Athens Insomnia Scale ( AIS ) is to assess subjective feelings about sleep.Using 0(no sleep disorders)-3(insomnia) rating form.
Change from Baseline of the ALT at 4 weeks | Baseline and Week 4
  Alanine aminotransferase, ALT in U/L
Change from Baseline of the AST at 4 weeks | Baseline and Week 4
  Aspartate aminotransferase, AST in U/L
Change from Baseline of the BUN at 4 weeks | Baseline and Week 4
  Blood urea nitrogen, BUN in mmol/L
Change from Baseline of the Scr at 4 weeks | Baseline and Week 4
  Serum creatinine, Scr in μmol/L
Genome-wide association study | Month 6
  Illumina HumanHap550-Duo BeadChips was used to perform the whole genome genotyping in deCODE genetics(Reykjavı'k, Iceland)
Item Patient Health Questionnaire ( PHQ-9 ) | Baseline and Week 4
  The PHQ-9 is a validated, self-reported questionaire aidding Auxiliary depression diagnosis and symptom severity assessment. Possible scores range from 0 (no depressive symptoms) to 27(major depression).
Change from Baseline in the score of Morningness-Eveningness Questionaire (MEQ) | Baseline and Week 4
  The MEQ is a validated, self-reported questionaire assessing personal chronotype in the recent period. Possible scores range from 16 (extreme eveningness) to 86 (extreme morningness). Change = (Week 4 Score - Baseline Score). Positive score change indicates a shift from eveningness to morningness.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No